CLINICAL TRIAL: NCT07295652
Title: Characterization of High-level Cognitive Impairments in Patients With Neuropsychiatric Disorders
Acronym: COGPSY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier St Anne (Other)
Collaborators: Institut du Cerveau et de la Moelle (ICM Institute) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D22-P009
Record Dates: First submitted 2025-06-13; First posted 2025-12-19 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Neurologic Disorders; Schizophrenia; Bipolar Disorder (BD); Depressive Disorder
Keywords: Cognitive dysfunction; Executive function; Metacognition; Motivation; Social cognition; Transdiagnostic approach; High-level cognition; Longitudinal cognitive changes; Cognitive profiling; Differential diagnosis
MeSH Terms: conditions — Nervous System Diseases; Schizophrenia; Bipolar Disorder; Depressive Disorder; Cognitive Dysfunction | interventions — Mental Status and Dementia Tests; Magnetoencephalography

STUDY DESIGN:
Intervention Model Description: This interventional study includes two distinct populations: patients with severe neuropsychiatric or neurological disorders, and healthy volunteers. All participants undergo the same cognitive assessments and evaluations. There is no randomization or allocation to different intervention arms; instead, all subjects receive the same intervention protocol for comparative purposes
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cognitive assessment (Experimental): Neuropsychological assessment assessing different cognitive dimensions (e.g., motivation and decision-making, metacognition, access to consciousness, Bayesian inference)
  Interventions: Behavioral: Cognitive assessment; Behavioral: Brain MRI (optional); Behavioral: Electroencephalography (optional); Behavioral: Magnetoencephalography (optional)

INTERVENTIONS:
Behavioral: Cognitive assessment — This intervention consists of computerized neuropsychological assessments designed to evaluate high-level cognitive impairments. The tests cover various cognitive dimensions including motivation, metacognition, conscious access, and Bayesian causal inference. These assessments are performed using computers or tablets, aiming to build a multidimensional cognitive atlas comparing patients with severe psychiatric and neurological conditions to healthy volunteers. The tests will be progressively optimized for usability and adapted to the specific difficulties faced by patients. For some participants, additional brain imaging (MRI without contrast, EEG, MEG) may be offered optionally to identify neural correlates of cognitive deficits.
Behavioral: Brain MRI (optional) — Brain MRI without contrast perform at one visit to identify neural correlates of cognitive deficits
Behavioral: Electroencephalography (optional) — Electroencephalography performed at one visit
Behavioral: Magnetoencephalography (optional) — Magnetoencephalography performed at one visit

SUMMARY:
Neuropsychiatric disorders are extremely common, severe, and disabling conditions. In the field of psychiatry, they notably include schizophrenia, mood disorders (depressive and bipolar disorders), autism spectrum or neurodevelopmental disorders, obsessive-compulsive disorder, eating disorders, and personality disorders. In the field of neurology, one can cite neurodegenerative diseases (such as Alzheimer's disease, but also frontotemporal dementia or Parkinson's disease, which often represent frequent and challenging differential diagnoses of psychiatric disorders), focal neurological lesions (notably strokes and tumors), or epilepsy.

Cognitive impairments are present in nearly all neuropsychiatric disorders and contribute significantly to disability.

While impairments in working memory and attention, executive functions, and social cognition have been relatively well studied, other cognitive domains remain largely unexplored in these populations. This is particularly the case for various aspects of motivation, metacognition, conscious access, or causal (Bayesian) inference.

Although these domains likely play an important role in prognosis, no consensus currently exists regarding the methods for evaluating these functions.

The main objective of this study is to define a multidimensional, transdiagnostic atlas of high-level cognitive impairments-both specific and shared-across severe psychiatric disorders (notably schizophrenia, depressive disorder, bipolar disorder, autism spectrum or neurodevelopmental disorders, and obsessive-compulsive disorder) and neurological disorders (notably neurodegenerative diseases, focal neurological lesions, and epilepsy), by comparing them to healthy volunteers.

The investigators also aim to investigate the progression of cognitive impairments over time, across different phases of illness (symptom stabilization or exacerbation) or therapeutic intervention, through longitudinal follow-up of patients being monitored within the recruiting center.

Finally, in a more exploratory manner, the investigators aim to investigate the neural correlates of the identified cognitive impairments.

DETAILED DESCRIPTION:
This study aims to construct a multidimensional, transdiagnostic atlas of high-level cognitive alterations across a range of severe neuropsychiatric conditions. These include schizophrenia, depressive disorders, bipolar disorder, autism spectrum or neurodevelopmental disorders, and obsessive-compulsive disorder, as well as neurological disorders such as neurodegenerative diseases, focal neurological lesions, and epilepsy. Cognitive performance in these groups will be compared to that of healthy volunteers in order to identify both disorder-specific and shared impairments.

Beyond this primary aim, the study seeks to refine and optimize the cognitive assessment tools used. Tests will be progressively adapted to be more ergonomic, shorter, and better suited for populations with neuropsychiatric conditions. This includes enhancing their intuitiveness, informativeness, and adaptability for digital platforms (e.g., tablet or mobile), while maintaining prior validation and calibration in healthy populations. The adaptation process will be informed by participant feedback and interim analysis.

The study will also examine how cognitive impairments evolve over time and with clinical changes, in participants undergoing psychiatric or neurological follow-up. Repeated cognitive evaluations will be scheduled in relation to clinical evolution, particularly before and after therapeutic interventions used in standard care, such as pharmacological treatment, non-invasive neurostimulation, psychotherapy, or psychoeducation.

In addition, the neural correlates of cognitive impairments will be explored using existing clinical brain imaging when available. Participants without prior imaging may be invited to undergo MRI scans, potentially including additional sequences such as DTI or functional MRI, without contrast administration. Complementary assessments using EEG or MEG may also be conducted, employing classical analyses such as event-related potentials and time-frequency analysis.

In some cases, causal inferences may be drawn by linking specific brain lesions in neurological patients to observed cognitive impairments. Finally, the study will explore whether selected cognitive tests could assist in differential diagnosis between psychiatric and neurological conditions, particularly neurodegenerative disorders.

This is a prospective, multicenter interventional study involving both healthy individuals and patients. It is classified as a minimal-risk, low-burden study and is designed to support the development of a comprehensive, comparative database of high-level cognitive dysfunctions across severe neuropsychiatric disorders.

ELIGIBILITY:
Inclusion Criteria:

For patients:

* Aged over 18 years
* Diagnosed with a psychiatric disorder according to ICD-10 by a psychiatrist (F10-F98) or diagnosed with a neurological disorder according to ICD-10 by a neurologist (G00-G99)
* Provided written informed consent
* Affiliated with a social security scheme

For healthy volunteers:

* Aged over 18 years
* Provided written informed consent
* Affiliated with a social security scheme

Exclusion Criteria:

For healthy volunteers:

* Current diagnosis of a psychiatric disorder according to ICD-10 (F20-F98) or current prescription of a psychotropic medication, or diagnosis of a neurological disorder according to ICD-10 (G00-G99)
* History of depression (F32)
* Substance use disorder (excluding tobacco)
* Neurological history (e.g., stroke, coma, epilepsy, neuroinflammatory or neurodegenerative disease) or identified cognitive disorder
* Inability to complete cognitive testing (e.g., due to motor or sensory impairment)

For participants undergoing MRI (without contrast agent):

* Presence of MRI contraindications: non-MRI-compatible pacemaker, heart valve, implant, or metallic foreign body
* Pregnancy at the time of MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-03-12 (Actual); Primary Completion 2039-03 (Estimated); Study Completion 2039-03 (Estimated)

PRIMARY OUTCOMES:
Performance scores on validated computerized neuropsychological tasks assessing high-level cognitive domains | Baseline, and up to one year after baseline
  Cognitive functions will be assessed using a battery of validated computerized neuropsychological tasks. The specific tasks will be selected and optimized for each target population, based on prior validation in healthy controls. Performance scores (e.g., accuracy, reaction time, decision-making indices) will be compared between patients with severe neuropsychiatric disorders and healthy volunteers.

SECONDARY OUTCOMES:
Optimization of performance scores on validated computerized neuropsychological tasks | Baseline, and up to one year after baseline
  A battery of validated computerized neuropsychological tasks will be progressively optimized based on participant feedback and interim analyses. The convergence of performance scores will be evaluated over multiple trials to refine the tests, ensuring suitability for populations with severe neuropsychiatric or neurological disorders.
Change from baseline in performance scores on validated computerized neuropsychological tasks | Baseline, and up to one year after baseline
  Changes in cognitive performance scores over time among patients undergoing standard clinical care, including therapeutic interventions. Cognitive evaluations will be repeated before and after major clinical events or treatment changes to assess cognitive stability or improvement
Structural and functional MRI | At MRI visit, between baseline and study completion (up to 10 years for patients; up to 1 year for healthy volunteers)
  Structural and functional MRI will be used to generate brain maps measuring gray matter volume (VBM), connectivity (DTI), and regional activation (fMRI). These MRI markers will be related to cognitive performance scores obtained during cognitive testing. Participation in MRI assessments is optional.
Electroencephalography (EEG) event-related potentials (ERP) during cognitive tasks | At EEG visits, from baseline through study completion (up to 10 years for patients; up to 1 year for healthy volunteers)
  EEG recordings will be performed during cognitive tasks. Event-related potentials (ERP) will be analyzed to investigate neurophysiological correlates of cognitive performance. These markers will be related to cognitive alterations in patients and compared across groups. Participation in EEG assessments is optional.
EEG time-frequency analyses during cognitive tasks | At EEG visits, from baseline through study completion (up to 10 years for patients; up to 1 year for healthy volunteers)
  EEG recordings will be performed during cognitive tasks. Time-frequency analyses will be used to investigate neurophysiological correlates of cognitive performance. These markers will be related to cognitive alterations in patients and compared across groups. Participation in EEG assessments is optional.
Magnetoencephalography (MEG) event-related potentials (ERP) during cognitive tasks | At MEG visits, from baseline through study completion (up to 10 years for patients; up to 1 year for healthy volunteers)
  MEG recordings will be performed during cognitive tasks. Event-related potentials (ERP) will be analyzed to investigate neurophysiological correlates of cognitive performance. These ERP markers will be related to cognitive alterations in patients and compared across groups. Participation in MEG assessments is optional.
MEG time-frequency analyses during cognitive tasks | At MEG visits, from baseline through study completion (up to 10 years for patients; up to 1 year for healthy volunteers)
  MEG recordings will be performed during cognitive tasks. Time-frequency analyses will be used to investigate neurophysiological correlates of cognitive performance. These markers will be related to cognitive alterations in patients and compared across groups. Participation in MEG assessments is optional.
Predictive capacity of cognitive performance scores for differential diagnosis | Baseline, and up to one year after baseline
  Validated cognitive performance tests will be used to evaluate patients longitudinally. The evolution of scores over time will be analyzed to determine the ability of these tests to discriminate between common differential diagnoses, such as frontotemporal dementia and depression. This outcome reflects the predictive capacity of cognitive tests for the final clinical diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Pierre BOURDILLON, Dr, Principal Investigator — Hôpital Fondation Adolphe de Rothschild
Locations (3):
- France (3):
  - Departement of Adult Psychiatry, GH Pitié Salpétrière, Paris
  - Groupe hospitalo-universitaire Paris Psychiatrie et Neurosciences, Paris
  - Hôpital Fondation Adolphe de Rothschild, Paris

IPD SHARING:
Plan to Share IPD: Yes
The data obtained from medical visits (clinical informations, cognitive data, medical imaging, and EEG/MEG recordings) will be kept, coded and archived for a period of two years after the last publication of the research results or until the final research report is signed. These can be used later for collaborative research (academic and/or industrial partners) in the European Union (EU) and/or abroad exclusively for scientific purposes.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data obtained from medical visits (clinical informations, cognitive data, medical imaging, and EEG/MEG recordings) will be kept, coded and archived for a period of two years after the last publication of the research results or until the final research report is signed.
Access Criteria: The data can be used for collaborative research (academic and/or industrial partners) in the European Union (EU) and/or abroad exclusively for scientific purposes. Any party must contact the sponsor, who has full property of the data.
  In case of requested transfer of the anonymized database resulting from this research abroad (outside the EU), the sponsor will request information regarding data storage and management, to make sure that the other party will be able to ensure a level of security equivalent to French or European Union law.